CLINICAL TRIAL: NCT02216747
Title: Treatment of Nephrotic Syndrome Relapse With Low Steroid Dose
Brief Title: Low Dose Steroids in the Treatment of Nephrotic Syndrome Relapse
Acronym: NS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Amit Dagan, DR. Amit Dagan, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC14 6413 CTIL
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Glomerular Disease
Keywords: Idiopathic Nephrotic syndrome relapse
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- prednisone 60 mg/meter square Body Surface Aera (Active Comparator): A - 60 mg Prednisone/meter square Boby Surface Area( 30 twice)/day until there are 3 days of undetected protein in urine and tapering down to 40 mg ,30 mg, 20 mg ,10 mg and 5 mg and end.
  Interventions: Drug: prednisone 60 mg/meter square Body Surface Area
- prednisone 45 mg/meter square BSA (Active Comparator): B- 45 mg prednisone / day until there are 3 days of undetected protein in urine and then 30 mg / day for two weeks and to 30,20,10,5 mg until treatment is ended.
  Interventions: Drug: prednisone 45 mg
- prednisone 30 mg/meter squer BSA (Active Comparator): C- treatment of twice daily prednisone 30 mg per day until there are 3 days of undetectible protein in urine and then tapering down to 20 ,10 ,5 until treatment is ended.
  Interventions: Drug: prednisone 30 mg

INTERVENTIONS:
Drug: prednisone 60 mg/meter square Body Surface Area — treatment with prednisone 60 mg /meter square Body Surface Area to compare to other arms
  Other Names: Danalon
  Arms: prednisone 60 mg/meter square Body Surface Aera
Drug: prednisone 45 mg — treatment with 45 mg prednisone to compare with other arms
  Other Names: Danalon
  Arms: prednisone 45 mg/meter square BSA
Drug: prednisone 30 mg — treatment with 30 mg prednisone to compare with other arms.
  Other Names: Danalon
  Arms: prednisone 30 mg/meter squer BSA

SUMMARY:
Background- Idiopathic Nephrotic syndrome is the common glomerular disease in childhood. conventional treatment is steroid treatment and nearly 90% response to this treatment well.

Response to this treatment is the most important prognostic factor and this patients has a benign disease course.

60-70% among patients that response to steroid treatment,will suffer a relapse of NS.repeated steroids courses can lead to serious adverse events in children such as low bone density,weight gain ,growth slow down ,elevated blood pressure and eye pressure.there is side effect corelation between steroid dose and treatment duration.

guidelines for steroid dose for NS relapse are not based on retrospective clinical research but only on Nephrologists and experts opinion.

Rational- What would be the optimal low dose steroids and the shortest time of treatment in Nephrotic syndrome relapse?

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome in children is the most common chronic glomerular disease. The first line of therapy is prednisone and about 90% of the patients will

response to this treatment. The course of the disease is characterized of

recurrent relapses and repeated prednisone therapy. While prednisone doses and

therapy duration in the disease diagnosis has been based on multiple prospective

studies, the dose and therapy duration in the relapses was never challenged in a

prospective control study.

To address this question we designed prospective 3 arm study to evaluate the

effective of exception steroid regiment to treat relapses versus lower doses.

The study population is children in the age 2-18 year old with steroid sensitive nephrotic syndrome.

After relapse will be diagnosed based on physical exam and urine tests, the

patients will randomize to receive prednisone doses that are 60/m2 or 45/ m2 or 30/ m2.

A measurement of time to obtain remission, duration of remission est. will be collected.

We plan to recruit 100 children in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Idiopathic nephrotic syndrome with a flair that needs steroids treatment.

Exclusion Criteria:

* Steroid resistance or treatment with Cyclosporin or Cellcept

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Nephrotic Syndrome Remission | 3 days
  Undetectable protein in urine for 3 days

SECONDARY OUTCOMES:
Remission duration | Weeks
  The number of weeks since the patient stopped steroids therapy and was in a complete remission.

OTHER OUTCOMES:
Edema | within 14 days
  A sign of treatment resistance or no response.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Dagan, Doctor, Principal Investigator — nephrology institute Shneider Children Hospital; Amit Dagan, Doctor, Principal Investigator — Schneider childrens Hospital Nephrology Institute
Locations (1):
- Shneider children Hospital Nephrology Institute, Petah Tikva, Israel

REFERENCES:
- [Derived] Hahn D, Samuel SM, Willis NS, Craig JC, Hodson EM. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD001533. doi: 10.1002/14651858.CD001533.pub7. PMID 39171624